CLINICAL TRIAL: NCT00368654
Title: An Open-Label Study to Evaluate Whether a Short-Term Course of Methotrexate in Psoriasis Patients Treated With Efalizumab is Safe and Increases Efficacy
Brief Title: Evaluate Whether Combination Therapy With Methotrexate and Raptiva in Psoriasis Patients is Safe and Increases Efficacy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200513613
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Results first posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Methotrexate; efalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A (Active Comparator): Monotherapy with Raptiva alone
  Interventions: Drug: Raptiva
- B (Experimental): Combination therapy with both Raptiva and Methotrexate
  Interventions: Drug: Methotrexate; Drug: Raptiva
- C (Experimental): Continue Raptiva, discontinue methotrexate
  Interventions: Drug: Raptiva
- D (Experimental): Continue combination therapy with both Raptiva and Methotrexate
  Interventions: Drug: Methotrexate; Drug: Raptiva

INTERVENTIONS:
Drug: Methotrexate — Initial dose 5 mg, then 15 mg per week
  Arms: B; D
Drug: Raptiva — Raptiva, initial dose 0.7 mg/kg, then 1.0 mg/kg
  Other Names: Efalizumab

SUMMARY:
To evaluate whether a short-term course of methotrexate in patients treated with efalizumab (Raptiva) increases efficacy. The secondary objectives of this study are 1) to evaluate the efficacy of Raptiva in maintaining the clinical improvement induced by short-term treatment with combination therapy of Raptiva and methotrexate 2) to evaluate the safety of short-term combination therapy of Raptiva and methotrexate.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate whether a short-term course of methotrexate in patients treated with efalizumab (Raptiva) increases efficacy. The secondary objectives of this study are 1) to evaluate the efficacy of Raptiva in maintaining the clinical improvement induced by short-term treatment with combination therapy of Raptiva and methotrexate 2) to evaluate the safety of short-term combination therapy of Raptiva and methotrexate.

The design of this study is to gain better control of the disease process while reducing potential toxicities by beginning treatment with Raptiva and adding methotrexate to those patients who do not improve significantly

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe plaque-type psoriasis
* A candidate for systemic therapy or phototherapy
* Not using prescription systemic therapies for psoriasis prior to starting the study
* Not using efalizumab within 3 months prior to starting the study

We are seeking adults who:

* Have moderate to severe plaque-type psoriasis
* Are generally healthy
* Are not hypersensitive to Raptiva® (efalizumab) or any of its components.
* Are not pregnant or lactating women

You will:

* Be interviewed and examined
* Have blood drawn
* Be injecting the study medication

Exclusion Criteria:

* Hypersensitivity to Raptiva or any of its components
* Pregnant or lactating women
* History of liver disease or abnormal liver enzymes
* History of chronic infection or malignancy
* History of significant hematologic abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chai Sue Lee, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical

RESULTS

PARTICIPANT FLOW:
Groups:
- A-Monotherapy With Raptiva Alone: Monotherapy with Raptiva alone
  Raptiva: Raptiva, initial dose 0.7 mg/kg, then 1.0 mg/kg
- B-Combination Therapy With Both Raptiva and Methotrexate: Combination therapy with both Raptiva and Methotrexate
  Methotrexate: Initial dose 5 mg, then 15 mg per week
  Raptiva: Raptiva, initial dose 0.7 mg/kg, then 1.0 mg/kg
- C-Continue Raptiva, Discontinue Methotrexate: Continue Raptiva, discontinue methotrexate
  Raptiva: Raptiva, initial dose 0.7 mg/kg, then 1.0 mg/kg
- D-Continue Combination Therapy With Both Raptiva and Methotrex: Continue combination therapy with both Raptiva and Methotrexate
  Methotrexate: Initial dose 5 mg, then 15 mg per week
  Raptiva: Raptiva, initial dose 0.7 mg/kg, then 1.0 mg/kg
Period: Overall Study
Arm/Group | A-Monotherapy With Raptiva Alone | B-Combination Therapy With Both Raptiva and Methotrexate | C-Continue Raptiva, Discontinue Methotrexate | D-Continue Combination Therapy With Both Raptiva and Methotrex
Started | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A-Monotherapy With Raptiva Alone | B-Combination Therapy With Both Raptiva and Methotrexate | C-Continue Raptiva, Discontinue Methotrexate | D-Continue Combination Therapy With Both Raptiva and Methotrex | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — data not collected | NA (NA) — data not collected | NA (NA) — data not collected | NA (NA) — data not collected | NA (NA) — data not collected
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — data not collected | NA — data not collected | NA — data not collected | NA — data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — data not collected | NA — data not collected | NA — data not collected | NA — data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: PASI -- Psoriasis Area and Severity Index
Description: (PASI) - given by numerical score, the index shows the severity of psoriasis.
Time Frame: 16 vs. 36 weeks, depending on study arm
Population: data not collected
Arm/Group | A-Monotherapy With Raptiva Alone | B-Combination Therapy With Both Raptiva and Methotrexate | C-Continue Raptiva, Discontinue Methotrexate | D-Continue Combination Therapy With Both Raptiva and Methotrex
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Adverse Events (AE)
Description: measured by whether or not AE was serious
Time Frame: 16 vs. 36 weeks, depending on study arm
Population: Data not collected
Arm/Group | A-Monotherapy With Raptiva Alone | B-Combination Therapy With Both Raptiva and Methotrexate | C-Continue Raptiva, Discontinue Methotrexate | D-Continue Combination Therapy With Both Raptiva and Methotrex
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | A-Monotherapy With Raptiva Alone | B-Combination Therapy With Both Raptiva and Methotrexate | C-Continue Raptiva, Discontinue Methotrexate | D-Continue Combination Therapy With Both Raptiva and Methotrex
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No